CLINICAL TRIAL: NCT04368910
Title: A Phase III Randomised, Double-blind, Double-dummy, Comparative Study to Assess the Safety and Efficacy of Pyronaridine Artesunate (180:60 mg) Versus Chloroquine (155 mg) in Children and Adult Patients in Korea With Acute P. Vivax Malaria
Brief Title: Safety and Efficacy of Pyronaridine Artesunate Vs Chloroquine in Children and Adult Patients With Acute Vivax Malaria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to slow recruitment the study was terminated prematurely by the Sponsor after 30 subjects had been included
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-C-008-07
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-11

CONDITIONS: Malaria
Keywords: Artemisinin-based combination therapy (ACT); Pyramax; Pyronaridine artesunate; Chloroquine; Children; Adults; Plasmodium vivax; Republic of Korea
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — pyronaridine tetraphosphate, artesunate drug combination; Chloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pyronaridine - artesunate (Experimental): Oral pyronaridine artesunate (180:60 mg tablets), plus chloroquine-placebo once a day for 3 consecutive days.
  For patients who complete the study up to Day 28 and who have normal G-6-PD activity, a 14-day course of primaquine (15 mg/day) shall be administered starting on Day 28, after all required assessments have been performed, to complete their radical cure. Patients who are deficient in G-6-PD and who complete the study up to Day 28 will be treated as per country policy.
  Interventions: Drug: Pyronaridine - artesunate
- Chloroquine (Active Comparator): Oral chloroquine (155 mg tablets), plus pyronaridine artesunate-placebo, once a day for 3 consecutive days.
  For patients who complete the study up to Day 28 and who have normal G-6-PD activity, a 14-day course of primaquine (15 mg/day) shall be administered starting on Day 28, after all required assessments have been performed, to complete their radical cure. Patients who are deficient in G-6-PD and who complete the study up to Day 28 will be treated as per country policy.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Pyronaridine - artesunate — Oral pyronaridine artesunate (180:60 mg tablets), plus chloroquine-placebo once a day for 3 consecutive days.
  Other Names: Pyramax
  Arms: Pyronaridine - artesunate
Drug: Chloroquine — Oral chloroquine (155 mg tablets), plus pyronaridine artesunate-placebo, once a day for 3 consecutive days.
  Arms: Chloroquine

SUMMARY:
The primary objective of this clinical study is to compare the efficacy and safety of the fixed combination of pyronaridine artesunate (180:60 mg) with that of standard chloroquine therapy in children and adults with acute, uncomplicated Plasmodium vivax (P. vivax) malaria

DETAILED DESCRIPTION:
This is a multi-centre, randomised, double-blind, double-dummy, parallel group, comparative trial. It is a Phase III study designed to meet the regulatory requirements for registration of pyronaridine artesunate (PA) in Korea. Chloroquine will be used as a comparator, which is recognized as an effective and well-tolerated anti-malarial therapy, and is standard blood-stage therapy for patients with P. vivax malaria in Korea. This study will be conducted in a total of 40 male and female children (≥20 kg body weight) and adult patients suffering from acute symptomatic uncomplicated P. vivax malaria recruited from study sites in Korea.

Patients will be randomised in a 1:1 ratio to receive either oral PA (180:60-mg tablets) plus chloroquine-placebo or oral chloroquine (155 mg tablets) plus PA-placebo, once a day for 3 consecutive days (Days 0, 1, and 2). For PA, posology will be based on body weight ranges, with patients receiving 1 to 4 tablets per day depending on their body weight. The actual dose range covered by this regimen is 7.2:2.4 mg/kg to 13.8:4.6 mg/kg per day, which has been shown to be effective and safe in Phase I and II studies. The chloroquine daily dose is 10 mg/kg on Days 0 and 1 and 5 mg/kg on Day 2 for children and 620 mg on Days 0 and 1 and 310 mg on Day 2 for adults.

Patients will be confined to the study facility for ≥4 days (Days 0, 1, 2, and 3) and remain near the study site for ≥7 days, or once fever and parasite clearance has been confirmed for ≥24 hours - whichever occurs later.

The primary efficacy end point for the study is the crude cure rate on Day 14. Scheduled follow-up visits will continue until completion of the study at Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

It is anticipated that the study results will be pooled with the results of study SP-C-006-06 entitled "A Phase III Comparative (Double-blind, Double-dummy) Randomized Multicentre Study to Assess the Safety & Efficacy of Oral Pyronaridine Artesunate (180:60 mg) Versus Chloroquine (155 mg) in Children & Adult Patients with Acute Vivax Malaria " for a formal non-inferiority analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 3 and 60 years, inclusive.
2. Body weight between 20 kg and 90 kg with no clinical evidence of severe malnutrition.
3. Presence of acute uncomplicated P. vivax mono-infection confirmed by:

   1. Fever, as defined by axillary/tympanic temperature ≥37.5°C or oral/rectal temperature ≥38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   2. Positive microscopy of P. vivax with parasite density ≥250/ μL of blood (including at least 50% of asexual parasites).
4. Written informed consent, in accordance with local practice, provided by patient and/or parent/guardian/spouse. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations.
5. Ability to swallow oral medication.
6. Ability and willingness to participate based on information given to patient or parent or guardian and access to health facility.

Exclusion Criteria:

1. Presence of a mixed Plasmodium infection.
2. Presence of other clinical condition requiring hospitalization.
3. Presence of significant anaemia, as defined by Hb <8 g/dL.
4. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTc interval greater than or equal to 450 msec), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including recent head trauma).
5. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine, chloroquine or artesunate or other artemisinins.
6. Known history of hypersensitivity, allergic or adverse reactions to chloroquine, primaquine and related agents.
7. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab).
8. Known seropositive HIV antibody.
9. Have received any antimalarial treatment in the preceding 2 weeks, as determined by history and, whenever feasible, by screening test.
10. Have received antibacterial with known antimalarial activity in the preceding 2 weeks.
11. Have received any investigational drug within the past 4 weeks.
12. Liver function tests (AST/ALT levels) >2.5 times the upper limit of normal range.
13. Known significant renal impairment as indicated by serum creatinine levels of >1.4 mg/dL.
14. Female patients of child-bearing potential must be neither pregnant (as demonstrated by a negative pregnancy test) nor lactating, and must be willing to take measures to not become pregnant during the study period.
15. Previous participation in the present clinical trial with pyronaridine artesunate.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09-06 (Actual); Primary Completion 2010-10-16 (Actual); Study Completion 2010-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Duparc, MD, Study Director — Medicine for Malaria Venture
Locations (2):
- South Korea (2):
  - Inje University Ilsan Paik Hospital, Goyang-si
  - Eulji General Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population: all randomized subjects (>12 years) who received any amount of study medication; subjects were analyzed as treated.
Groups:
- Pyronaridine - Artesunate: Oral pyronaridine artesunate (180:60 mg tablets), plus chloroquine-placebo once a day for 3 consecutive days.
  For patients who complete the study up to Day 28 and who have normal G-6-PD activity, a 14-day course of primaquine (15 mg/day) shall be administered starting on Day 28, after all required assessments have been performed, to complete their radical cure. Patients who are deficient in G-6-PD and who complete the study up to Day 28 will be treated as per country policy.
  Pyronaridine - artesunate: Oral pyronaridine artesunate (180:60 mg tablets), plus chloroquine-placebo once a day for 3 consecutive days.
- Chloroquine: Oral chloroquine (155 mg tablets), plus pyronaridine artesunate-placebo, once a day for 3 consecutive days.
  For patients who complete the study up to Day 28 and who have normal G-6-PD activity, a 14-day course of primaquine (15 mg/day) shall be administered starting on Day 28, after all required assessments have been performed, to complete their radical cure. Patients who are deficient in G-6-PD and who complete the study up to Day 28 will be treated as per country policy.
  Chloroquine: Oral chloroquine (155 mg tablets), plus pyronaridine artesunate-placebo, once a day for 3 consecutive days.
- Total: Total of all reporting groups
Arm/Group | Pyronaridine - Artesunate | Chloroquine | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (14.03) | 42.3 (11.79) | 40.3 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Oriental | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Crude Cure Rate on Day 14
Description: Percentage of subjects with crude cure rate at Day 14, defined as absence of parasitaemia on Day 14, irrespective of body temperature without previously meeting any of the criteria of treatment failure
Time Frame: Day 14
Population: Efficacy evaluable population: completed a full course of study medication, did not miss a dose, did not use a concomitant medication that may have interfered with the treatment outcome up to D14, did not have a concomitant disease which may have interfered with the classification of the treatment outcome, did not have major protocol deviations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
percentage of participants | 100 [75.3 to 100.0] | 100 [78.2 to 100.0]

2. Secondary Outcome: Crude Cure Rate on Day 28
Description: Percentage of subjects with crude cure rate at Day 28, defined as absence of parasitaemia on Day 28, irrespective of body temperature without previously meeting any of the criteria of treatment failure
Time Frame: Day 28
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
percentage of participants | 100 [75.3 to 100.0] | 100 [78.2 to 100.0]

3. Secondary Outcome: Parasite Clearance Time (PCT)
Description: Parasite clearance time is defined as the time from first dosing to the time of first blood draw with parasite clearance. Parasite clearance was defined as zero presence of asexual parasites for 2 consecutive negative readings taken between 7 and 25 hours apart
Time Frame: Days 0, 3, 7, 14, 21, 28, 35, and 42 (or on any other day if the subject spontaneously returned within the 42-day period)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
hours | 32.0 [24.0 to 40.0] | 63.9 [55.9 to 160.8]

4. Secondary Outcome: Fever Clearance Time (FCT)
Description: Fever clearance time is defined as the time from first dosing to the first normal reading of temperature for 2 consecutive normal temperature readings taken between 7 and 25 hours apart
Time Frame: Day 0 and every 8 hours over ≥72 hours following first study drug administration or temperature normalization for ≥2 readings between 7 and 25 hours apart, then at each visit (Days 7, 14, 28 and 42)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
hours | 16.0 [15.9 to 24.0] | 31.9 [23.5 to 39.8]

5. Secondary Outcome: Percentage of Patients Who Had Cleared Parasite on Days 1, 2, and 3
Description: Parasite clearance is defined as at least 2 consecutive negative smears for asexual parasites obtained within an interval of 7 to 25 hours post-dosing
Time Frame: Days 1, 2, and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
percentage of participants
  Day 1 (24h after first dose) | 30.8 [5.7 to 55.9] | 0.0 [0.0 to 0.0]
  Day 2 (48h after first dose) | 92.3 [77.8 to 100.0] | 26.7 [4.3 to 49.0]
  Day 3 (72h after first dose) | 100.0 [100.0 to 100.0] | 60.0 [35.2 to 84.8]

6. Secondary Outcome: Percentage of Patients Who Had Cleared Fever on Days 1, 2, and 3
Description: Fever clearance is defined as at least 2 consecutive normal body temperature measurements (<37.5 C axillary/tympanic or <38.0 C oral/rectal) obtained within an interval of 7 to 25 hours postdosing
Time Frame: Days 1, 2, and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
percentage of participants
  Clearance rate (%) at Day 1 (24h after first dose) | 76.9 [54.0 to 99.8] | 41.7 [13.8 to 69.6]
  Clearance rate (%) at Day 2 (48h after first dose) | 92.3 [77.8 to 100.0] | 91.7 [76.0 to 100.0]
  Clearance rate (%) at Day 3 (72h after first dose) | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

7. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of Participants with AEs, including clinically significant laboratory results, electrocardiogram (ECG), vital signs or physical examination abnormalities
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study
Population: Safety population, consisting of all randomised subjects who received any amount of study medication; subjects were analysed as treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 15 | 15
Participants
  Nr subj. with ≥1 AE | 10 | 10
  Nr subj. with ≥1 treatment-related AE | 7 | 9
  Nr subj. with ≥1 SAE | 0 | 0
  Nr subj. with ≥1 treatment-related SAE | 0 | 0
  Nr subj. with ≥1 severe or life-threatening AE | 0 | 2
  Nr subj. with ≥1 AE leading to death | 0 | 0
  Nr subj. with≥1 AE leading to drug discontinuation | 0 | 0
  Nr subj. with ≥1 AE leading to study withdrawal | 0 | 0

8. Other Pre Specified Outcome: Crude Cure Rate on Day 42
Description: Proportion of subjects with crude cure rate at Day 42, defined as absence of parasitaemia on Day 42, irrespective of body temperature without previously meeting any of the criteria of treatment failure
Time Frame: Day 42
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Pyronaridine - Artesunate | Chloroquine
Number analyzed (Participants) | 13 | 15
percentage of subjects | 100 [75.3 to 100.0] | 100 [78.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study
Arm/Group | Pyronaridine - Artesunate | Chloroquine
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 10/15 | 10/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyronaridine - Artesunate (N=15) | Chloroquine (N=15)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Drug-related AE
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) — Drug-related AE
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) — Drug-related AE
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) — Drug (PA)-related AE
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Drug-related AE
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Drug-related AE
Fatigue (General disorders) | 1 (1) | 1 (1) — Drug (PA)-related AE
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (2) — Drug-related AE
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1) — Drug-related AE
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) — Drug-related AE
Haematocrit decreased (Investigations) | 1 (1) | 0 (0) — Drug-related AE
Platelet count decreased (Investigations) | 1 (1) | 0 (0) — Drug-related AE
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) — Drug-related AE
White blood cell count increased (Investigations) | 1 (1) | 0 (0) — Drug-related AE
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) — Drug-related AE
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 1 (1) — Drug-related AE
Transaminases increased (Investigations) | 0 (0) | 1 (1) — Drug-related AE
Weight decreased (Investigations) | 0 (0) | 1 (1) — Drug-related AE
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Drug-related AE
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) — Drug-related AE
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Drug-related AE
Hypotension (Vascular disorders) | 0 (0) | 1 (1) — Drug-related AE

LIMITATIONS AND CAVEATS:
Due to slow recruitment the study was terminated prematurely by the Sponsor after 30 subjects (of the 40 planned) had been included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No